CLINICAL TRIAL: NCT06349746
Title: The Addition of Cervical Unilateral Antero-posterior Mobilization and Thoracic Central Postro-anterior Mobilization to Selected Therapeutic Exercise Program in Treatment of Shoulder Impingement Syndrome: A Randomized Clinical Trial
Brief Title: Cervical Unilateral Antero-posterior Mobilization and Thoracic Central Postro-anterior Mobilization in Treatment of Shoulder Impingement Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Chinese University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Noha Elserty, Assistant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: collage of physical therapy
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: this study will be conducted to compare one group receiving selected therapeutic exercises and other group recieve cervical and thoracic mobilization added to selected therapeutic exercise Program on pain intensity, Pain-free shoulder flexion and scaption active ROM, muscle strength of external rotator and abductors, shoulder functional status in patients with Shoulder Impingement Syndrome.
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and outcomes assessor will be masked about the grouping of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercises (Active Comparator): a specific therapeutic exercise program consisted of stretching exercises for posterior capsule and progressive resistance exercises for rotator cuff and scapula stabilizer and home exercise
  Interventions: Other: therapeutic exercises
- cervical and thoracic mobilization (Active Comparator): cervical unilateral antero-posterior mobilization and thoracic central postro-anterior mobilization added to therapeutic exercises
  Interventions: Other: mobilization exercise

INTERVENTIONS:
Other: therapeutic exercises — stretching exercise to posterior capsule and progressive resistance exercise for rotator cuff and scapula stabilizer and home exercise 3 sessions per week for 6 week.
  Arms: Therapeutic exercises
Other: mobilization exercise — cervical unilateral antero-posterior mobilization and thoracic central postro-anterior mobilization
  Arms: cervical and thoracic mobilization

SUMMARY:
Shoulder impingement syndrome (SIS) is a complex, multi-factorial problem that is treated with a variety of different conservative options. The conservative option that has shown effectiveness is manual therapy of the cervical and thoracic spine

DETAILED DESCRIPTION:
This study will be conducted to answer the following question:

What is the effect of adding cervical and thoracic mobilization to selected therapeutic exercise Program on pain intensity, Pain-free shoulder flexion and scaption active ROM, muscle strength of external rotator and abductors, shoulder functional status in patients with Shoulder Impingement Syndrome

ELIGIBILITY:
Inclusion Criteria:

* • patients who had received at least two positive signs on their Neer sign, Hawkins sign, supraspinatus test, apprehension test, and relocation test

  * Patients report pain on elevating the arm between 70 ° and 120 ° (the "painful arc"), on forced movement above the head, and when lying on the affected side

Exclusion Criteria:

* • cervical radiculopathy

  * a history of shoulder surgery
  * corticosteroid injection within the past month
  * Subjects who had received physical therapy treatment for their shoulder within the past three months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
pain intensity | pre intervention and after 6 weeks of intervention
  pain intensity will be measured by visual analogue scale
shoulder flexion and abduction range of motion | pre intervention and after 6 weeks of intervention
  measurement of shoulder flexion and abduction range of motion applied by using digital goniometer
muscle strength | pre intervention and after 6 weeks of intervention
  shoulder flexors and external rotators muscle strength will be measured by dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Noha Elserty, Principal Investigator — Benha University